CLINICAL TRIAL: NCT03235635
Title: Metagenome Analysis of Intestinal Microbiome in Mortality and Morbidity of Preterm Infants
Brief Title: Metagenomic Analysis of Gut Microbiome in Preterm
Acronym: MAGMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Byoungkook Lee, assistant professor, Wonju Severance Christian Hospital
Other Study IDs: microbiome in nicu
Record Dates: First submitted 2017-07-17; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Microbial Colonization; Microbial Superinvasion; Microbial Substitution; Newborn Morbidity
Keywords: microbiome; preterm; newborn; gut microbiome; allergic predisposition
MeSH Terms: conditions — Communicable Diseases; Superinfection; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — extraction microbiome DNA from stool of newborns
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preterm: newborn infants were born with a gestational age of less than 32 weeks
- Late preterm: newborn infants were born with a gestational age of greater than 32 weeks and less than 36 weeks
- full-term: newborn infants were born with a gestational age of greater than or equal to 37 weeks

SUMMARY:
This is single center study. The investigators will try to know that relationships between intestinal microbiome and mortality in preterm infants and what relationships is between intestinal microbiome in preterm infants and morbidity, mortality.

DETAILED DESCRIPTION:
Microbiome is the collection of all the microorganisms living in association with the human body which are consist of eukaryotes, archaea, bacteria and viruses. Microbiome in an average human body number are ten times more than human cells and have about 1000 more genes than are present in the human genome. There are symbiotic relationships between human and microbiome. If investigators are able to know about relationships between newborn and intestinal microbiome, mortality and morbidity in preterm infants may be improved. The investigators will collect the first and weekly stool of participants and analyze DNA of microbiome thorough Metagenomic anlysis. The results between 3 groups(preterm, late preterm and full-term infants) will be compared. The investigators expect that a mean distribution of intestinal microbiome in newborns(preterm, late preterm and full-term) is defined and that relationships between mortality, morbidity and intestinal microbiome.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants who were born at gestational age of less than 36 weeks from approval date to Feb 28th 2019
* full-term infants who were born at gestational age of greater than 37 weeks from approval date to Feb 28th 2019

Exclusion Criteria:

* newborns with congenital anomaly
* newborns with genetic syndrome
* newborns without consent of parents

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborn infants who were born and admitted on neonatal intensive care unit of Wonju Severance Christian Hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Intestinal microbiome | for 2 years
  The distribution rate of intestinal microbiome of stool by K-mer based taxonomic assignment which is one of the analysis in result of metagenomics in each infants

SECONDARY OUTCOMES:
Full Enteral feeding in preterm infants | for 2 years
  Days to accomplish a full-enteral feeding in each infants
Growth rate | for 2 years
  Days to reach 2 kg of body weight in each infants
Mortality | for 2 years
  Number of patients who died in neonatal intensive care unit.
Morbidity | for 2 years
  Number of patients who had a complication of preterm infants(e.g. necrotizing enterocolitis, bronchopulmonary dysplasia) or were died in neonatal intensive care unit.
Allergic predisposition | for 2 years
  Number of patients who were developed a allergic predisposition at 6 month of postnatal age.

CONTACTS AND LOCATIONS:
Overall Officials: Byoungkook Lee, Study Chair — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol
Time Frame: starting from august 2017 until February 2019
Access Criteria: neonatology pediatrics infections

REFERENCES:
- [Result] Rautava S. Microbial Composition of the Initial Colonization of Newborns. Nestle Nutr Inst Workshop Ser. 2017;88:11-21. doi: 10.1159/000455209. Epub 2017 Mar 27. PMID 28346920
- [Result] Butel MJ, Suau A, Campeotto F, Magne F, Aires J, Ferraris L, Kalach N, Leroux B, Dupont C. Conditions of bifidobacterial colonization in preterm infants: a prospective analysis. J Pediatr Gastroenterol Nutr. 2007 May;44(5):577-82. doi: 10.1097/MPG.0b013e3180406b20. PMID 17460489
- [Result] Turnbaugh PJ, Ley RE, Hamady M, Fraser-Liggett CM, Knight R, Gordon JI. The human microbiome project. Nature. 2007 Oct 18;449(7164):804-10. doi: 10.1038/nature06244. PMID 17943116
- [Result] Jacquot A, Neveu D, Aujoulat F, Mercier G, Marchandin H, Jumas-Bilak E, Picaud JC. Dynamics and clinical evolution of bacterial gut microflora in extremely premature patients. J Pediatr. 2011 Mar;158(3):390-6. doi: 10.1016/j.jpeds.2010.09.007. Epub 2010 Oct 18. PMID 20961563
- [Result] Arboleya S, Binetti A, Salazar N, Fernandez N, Solis G, Hernandez-Barranco A, Margolles A, de Los Reyes-Gavilan CG, Gueimonde M. Establishment and development of intestinal microbiota in preterm neonates. FEMS Microbiol Ecol. 2012 Mar;79(3):763-72. doi: 10.1111/j.1574-6941.2011.01261.x. Epub 2011 Dec 15. PMID 22126419
- [Result] Johnson CL, Versalovic J. The human microbiome and its potential importance to pediatrics. Pediatrics. 2012 May;129(5):950-60. doi: 10.1542/peds.2011-2736. Epub 2012 Apr 2. PMID 22473366
- [Result] McElroy SJ, Weitkamp JH. Innate Immunity in the Small Intestine of the Preterm Infant. Neoreviews. 2011 Sep 1;12(9):e517-e526. doi: 10.1542/neo.12-9-e517. PMID 22639551
- [Result] Groer MW, Luciano AA, Dishaw LJ, Ashmeade TL, Miller E, Gilbert JA. Development of the preterm infant gut microbiome: a research priority. Microbiome. 2014 Oct 13;2:38. doi: 10.1186/2049-2618-2-38. eCollection 2014. PMID 25332768